CLINICAL TRIAL: NCT06371768
Title: Symptom Management and Transitioning to Engagement With Post-treatment Care for Adolescent and Young Adult Cancer Survivors
Acronym: AYA STEPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00115400; 5R37CA283353-02 (NIH)
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cancer; Breast Cancer; Colorectal Cancer; Sarcoma; Lymphoma; Testicular Cancer
Keywords: Cancer; Young Adult; Behavioral Symptom Management
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Sarcoma; Lymphoma; Testicular Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Control (Active Comparator): The education control condition will match AYA STEPS in delivery format [videoconferencing, web-based platform, frequency (biweekly sessions)], and session number (six) and length.
  Interventions: Behavioral: AYA Educational Information
- AYA STEPS (Experimental): Participants will receive the AYA STEPS digital health intervention, which includes six sessions delivered remotely (i.e., videoconferencing) by a clinical psychologist with intervention content accessed using a web-based platform.
  Interventions: Behavioral: AYA STEPS

INTERVENTIONS:
Behavioral: AYA Educational Information — AYA-specific educational information is delivered using video conferencing by a clinical psychologist over six sessions. Participants will receive a written manual providing tips for engaging with educational content as well as access to a website specific to the control arm, which will provide written, video, and pictorial information.
  Arms: Education Control
Behavioral: AYA STEPS — The intervention provides cognitive-behavioral and patient activation theory-based skills designed to enhance AYA survivors' abilities to manage their high symptom burden and engage in follow-up health care. Sessions with the psychologist will focus on enhancing participants' abilities to apply intervention skills and engage in the AYA STEPS digital health intervention using motivational interviewing, goal setting, and problem-solving techniques. Participants will complete the six sessions over the 12 weeks of the AYA STEPS intervention.
  Arms: AYA STEPS

SUMMARY:
The purpose of this study is to determine the effectiveness of a digital health program called AYA STEPS, which is designed to help adolescent and young adult (AYA) cancer survivors manage symptoms and engage in recommended follow-up care.

DETAILED DESCRIPTION:
The investigators have developed an accessible digital health intervention, AYA STEPS (Symptom Management and Transitioning to Engagement with Post-Treatment Care for AYA Survivors), designed to enhance adolescent and young adult (AYA) cancer survivors' abilities to manage their high symptom burden and engage in follow-up health care. Informed by the Obesity-Related Behavioral Intervention Trials (ORBIT) Model of intervention development, AYA STEPS has been systematically and rigorously developed and refined through the PI's prior work (K08CA245107). AYA STEPS is organized into six remotely delivered sessions providing cognitive-behavioral and patient activation theory-based skills expected to lead to lower symptom burden and increased health care engagement by improving AYAs' self-efficacy for symptom management and activation. The investigators propose a randomized controlled trial to examine the efficacy of AYA STEPS compared to AYA educational information for improving symptom burden and health care engagement for AYA survivors (N=260) who received cancer care in diverse health care settings (i.e., rural, urban, medically underserved areas) across North Carolina. Self-efficacy and patient activation will be examined as mediators of intervention effects. The planned study has the potential to produce clinically impactful health benefits for an underserved and understudied group of cancer survivors who have significant symptom burden, experience barriers to care engagement, and have limited access to AYA-specific behavioral interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with one of the following cancers: 1) stage I-III breast cancer; 2) stage I-III colorectal cancer; 3) stage I-III sarcoma; 4) stage I-III Hodgkin or non-Hodgkin lymphoma; or 5) stage I-II testicular cancer
* treated with curative intent and off therapy (with the exception of endocrine/hormonal therapy or oral targeted therapies used to prevent disease recurrence or progression) for the last three months
* 1 to 5 years post-diagnosis
* Able to speak and read English
* Able to give informed consent

Exclusion Criteria:

* moderate or severe cognitive impairment
* severe untreated mental illness (e.g., schizophrenia, substance use disorder) that would interfere with providing meaningful consent/study participation

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Pain severity and interference as measured by Brief Pain Inventory | Baseline, 3 Months, 6 Months, 12 Months
  The Brief Pain Inventory will be used to assess pain severity and interference from pain across important life domains (e.g., general activity, work, relations with others). This measures includes a body map on which the patient can mark the location(s) in which they are experiencing pain, as well as 8 questions on a scale of 0 to 10 with higher scores indicating worse pain severity or pain interference.
Fatigue as measured by PROMIS Fatigue Scale | Baseline, 3 Months, 6 Months, 12 Months
  Fatigue will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Fatigue Scale, a 6-item self-report measure of fatigue. Participants are asked to think about the last week when responding to each item (e.g., "In the past 7 days, how run-down did you feel, on average?"), providing ratings on a scale from "not at all" (1) to "very much" (5).
Emotional distress as measured by PROMIS Depression Short Form | Baseline, 3 Months, 6 Months, 12 Months
  Depressive symptoms will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Short Form, an 8-item measure assessing symptoms of depression in the last week. Responses are on a 5-point scale from "never" (1) to "always" (5).
Emotional distress as measured by PROMIS Anxiety Short Form | Baseline, 3 Months, 6 Months, 12 Months
  Symptoms of Anxiety will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form, an 8-item measure assessing symptoms of anxiety in the last week. Responses are on a 5-point scale from "never" (1) to "always" (5).
Symptom interference as measured by MD Anderson Symptom Inventory (MDASI) Symptom Interference | Baseline, 3 Months, 6 Months, 12 Months
  The MDASI will be used to assess interference of symptoms in daily living (e.g., working, relations with other people, enjoyment of life) over the past month. The MDASI asks patients to rate the severity of 13 symptoms found frequently in patients with various cancers and treatment types on a scale from 0 (symptom "not present") to 10 (symptom "as bad as you can imagine"). This measure also includes 6 questions asking patients to rate the level of symptom interference in six domains (e.g., general activity, mood) on a scale from 0 (did not interfere) to 10 (interfered completely).
Health care engagement as measured by Patient Participation Questionnaire | Baseline, 3 Months, 6 Months, 12 Months
  The Patient Participation Questionnaire will be used to assess participants' health care participation and associated domains (i.e., receipt of information, communication, perceptions of their relationship with the medical team). Participants are asked to indicate their agreement with 17 items related to health care engagement on a 4 point scale: "to a great extent," "to some extent," "to a lesser extent," or "not at all." An additional item asks patients about their overall assessment of their involvement in their healthcare.
Patient self-assessment of communication competency with health care providers as measured by Medical Communication Competence Scale (MCCS) patient subscale | Baseline, 3 Months, 6 Months, 12 Months
  The MCCS patient subscale will be used to assess survivors' perceptions of their competency for communicating and participating in health care. The patient subscale includes 39 items on a scale of 1 to 7, with higher scores reflecting self-perception of better medical communication competence.

SECONDARY OUTCOMES:
Patient self-efficacy for chronic disease coping as measured by Self-Efficacy for Managing Chronic Illness Scale | Baseline, 3 Months, 6 Months, 12 Months
  The 6-item Self-Efficacy for Managing Chronic Illness Scale will be used to assess participants' current confidence in their ability to prevent symptoms (e.g., pain, fatigue, distress) from interfering with life. Responses are on a 10-point scale from "not at all confident" (1) to "totally confident" (10).
Patient activation as measured by Patient Activation Measure (PAM) | Baseline, 3 Months, 6 Months, 12 Months
  The PAM is a 13-item measure used to assess survivors' knowledge, skills, and confidence that are central to managing their health and health care. Patients are asked to rate their agreement with statements about their health and health care on a 4 point scale from "strongly disagree" to "strongly agree." From these response a total PAM score is calculated on a scale of 0-100, with higher scores indicating higher levels of activation.
Patient self-efficacy for managing chronic conditions as measured by the PROMIS Self-Efficacy for Managing Symptoms Short Form | Baseline, 3 Months, 6 Months, 12 Months
  The 4-item PROMIS Self-Efficacy for Managing Symptoms will be used to assess participants' confidence in their ability to manage symptoms (e.g. during daily activities, in a public place). Items are scored on a 5-point Likert scale, with higher scores indicating greater confidence.
General patient self-efficacy as measured by the PROMIS General Self-Efficacy Short Form | Baseline, 3 Months, 6 Months, 12 Months
  The 4-item PROMIS General Self-Efficacy will be used to assess participants' general confidence in their abilities (e.g., to solve problems and persist toward goals). Items are scored on a 5-point Likert scale, with higher scores indicating greater confidence.

OTHER OUTCOMES:
Health care utilization: Chart Review | 12 Months
  Health care utilization in the time since study enrollment will be assessed via review of participants' medical records to examine participants' receipt of general health screenings, cancer-related screenings, and follow-up care for late effects, in accordance with the 2024 National Comprehensive Cancer Network (NCCN) Adolescent and Young Adult (AYA) Guidelines.
Area Deprivation Index (ADI) | Baseline
  The ADI will be calculated using participants home mailing addresses. The ADI is an indexed composite of 17 variables related to social determinants of health from the United States Census and American Community Survey that captures socioeconomic disadvantage at the census block group level. The index is reported as a percentile from 0% to 100%, with higher scores indicating higher levels of deprivation.
Health-care utilization: Self-report | Baseline, 3 Months, 6 Months, 12 Months
  Participants' self-reports of their health care utilization since study enrollment will be collected to enhance the study team's ability to obtain chart review data.
Health literacy as measured by Medical Term Recognition Test (METER) | Baseline
  The METER will be used to assess health literacy. Participants are asked to review a list of 40 words and check off those that they recognize as actual words.
Participant experiences of discrimination as measured by Everyday Discrimination Scale-Short Form | Baseline
  The Everyday Discrimination Scale-Short Form is a 5-item scale that assesses participants' subjective experiences of daily discrimination, with patients indicating the frequency of discrimination experiences on a 6-point scale from "never" to "almost everyday." Patients who respond that they have experienced discrimination more frequently than "never" are asked what they think is the main reason(s) they experience(d) discrimination (e.g. ancestry, gender, race).
Participant evaluation of study mobile application as measured by User Version of the Mobile Application Rating Scale (uMARs) | 3 Months
  The 20-item uMARs will be adapted to obtain participants' evaluation of the AYA STEPS digital health platform and the AYA Educational Information website. Participants are asked to respond to questions regarding the quality of the mobile application on a 5-point scale from "inadequate" (1) to "excellent" (5). A total quality score is calculated as the mean of four objective quality subscales (engagement, functionality, aesthetics, and information quality). The uMARs also includes a subjective quality subscale.
Symptom interference as measured by the Illness Intrusiveness Rating Scale | Baseline, 3 Months, 6 Months, 12 Months
  The Illness Intrusiveness Rating Scale (IIRS) is a 13-item scale that assesses symptom interference across multiple life domains on a scale from 1 to 7, with higher scores indicating increased illness intrusiveness. The IIRS may be given a total sum score, or mean scores across three subscales: relationships and personal development, intimacy, and instrumental.
Satisfaction with Treatment and Interventionist as measured by the Satisfaction with Therapy and Therapist Scale-Revised (STTS-R) | 3 Months
  Participants will complete the 13-item Satisfaction with Therapy and Therapist Scale-Revised specific to the interventionists delivering either AYA STEPS or AYA Educational Information. The first 12 items ask participants to rate their agreement with statements related to intervention satisfaction on a 5-point scale ranging from "strongly disagree" (1) to "strongly agree" (5). The 13th item asks "How much did the intervention help with your symptoms?" with 5 answer choices ranging from "made things a lot better" to "made things a lot worse."
Web-based Portal Use as measured by total time using portal in minutes | Continuous (Baseline to 12 Months)
  The AYA STEPS web-based portal and AYA Education Information website will track overall participant usage and content access for each of the respective sessions. The investigators will examine time spent accessing session content and time spent engaging in and completing home practice assignments.
Emotional support as measured by the PROMIS Emotional Support Short Form | Baseline, 3 Months, 6 Months, 12 Months
  Emotional support will be assessed using the Patient-Reported Outcomes Measurement Information System (PROMIS) Emotional Support Short Form, a 6-item measure assessing patients' perceived emotional support. Responses are on a 5-point scale from "never" (1) to "always" (5).
Role functioning as measured by the 7-item role functioning subscale of the Functional Assessment of Cancer Therapy - General | Baseline, 3 Months, 6 Months, 12 Months
  The 7-item functional well-being subscale of the Functional Assessment of Cancer Therapy - General (FACT-G) will assess the impact of cancer and cancer therapy on role functioning by evaluating participants' agreement with statements assessing functional well-being on a scale of 0 ("Not at all") to 4 ("Very much"). Higher scores indicate greater functional well-being.
Spiritual well-being as measured by the Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Scale | Baseline, 3 Months, 6 Months, 12 Months
  The 12-item Functional Assessment of Chronic Illness Therapy Spiritual Well-Being Scale assesses spiritual well-being among patients with cancer. Participants report agreement with 12 statements assessing spiritual well-being on a scale of 0 ("Not at all") to 4 ("Very much"), with higher scores indicating greater spiritual well-being.
Patient congruence of behaviors with values as measured by the Valuing Questionnaire | Baseline, 3 Months, 6 Months, 12 Months
  The 10-item Valuing Questionnaire assesses congruence of behaviors with values by asking participants to rate their agreement with statements reflecting valued living on a scale of 0 ("Not at all true") to 6 ("Completely true"). Higher scores indicate higher congruence of behaviors with values.
Psychological flexibility as measured by the Acceptance and Action Questionnaire for Cancer | Baseline, 3 Months, 6 Months, 12 Months
  The 18-item Acceptance and Action Questionnaire for Cancer (AAQ-C) assesses psychological flexibility by asking participants to rate their agreement with 18 statements evaluating their experiences as cancer survivors, on a scale of 1 ("Never true") to 7 ("Always true"). Lower scores indicate greater psychological flexibility.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
It is the investigators' intention to make all data generated from this proposal freely available after it is de-identified. All direct respondent identifiers (e.g., names and addresses) will be removed and maintained in a secure file for future contact purposes. Respondent identifiers will not be shared. All other scientific data (scale composites) will be both preserved and shared. The following data will be preserved and shared: patient-reported data from study assessments, intervention utilization data collected via the study websites, healthcare utilization data collected from the health record, socio-demographic and medical data collected via patient report and health record, and scores on social determinant of health assessments (e.g., Area Deprivation Index). The investigators will make every effort to provide raw data in a non-proprietary format wherever possible to enhance reproducibility.